CLINICAL TRIAL: NCT01346423
Title: Is Interdisciplinary Intervention for Patients Sicklisted With Musculoskeletal Pain More Effective in Helping Patients Back to Work Than Than The Less Resource Demanding Brief Intervention Method?
Brief Title: Interdisciplinary Intervention Versus Brief Intervention for Patients With Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150160
Record Dates: First submitted 2011-04-14; First posted 2011-05-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2011-03

CONDITIONS: Musculoskeletal Diseases
Keywords: Sick leave; musculoskeletal pain; return to work; multidisciplinary intervention; randomised controlled trial
MeSH Terms: conditions — Musculoskeletal Diseases; Musculoskeletal Pain | interventions — Control Groups; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Treatment team with a physician, a physiotherapist, a social service worker. The main goal for the team is to make a survey of the patient's situation, in which the biomedical tradition to make a diagnosis is replaced by a disability diagnosis, with systematically identification of barriers for return to work. The patient meets at the outpatient clinic three times; at baseline, after 2 weeks and after 3 months. One year after baseline the patient has a telephone-follow-up. At baseline, the patient and the team works out a rehabilitation plan and in this process a new visual, educational tool is central.
  Interventions: Behavioral: Interdisciplinary intervention
- Controll group (Active Comparator): The brief intervention is a standardized intervention based on the studies by Indahl and Hagen. Therapist treatment manuals will be written for the intervention. The essential features are interview and examination by a specialist in physical medicine and rehabilitation. Patients will be given time to express their concerns and problems in daily activities. Unless symptoms and clinical findings indicate some serious disease, the patients will be informed about the good prognosis, and the importance of staying active to avoid development of muscle dysfunction.
  Interventions: Behavioral: Control Group, Brief Intervention

INTERVENTIONS:
Behavioral: Interdisciplinary intervention — Interdisciplinary collaboration deals with tasks often complex which require different skills to make a wide assessment.In this study the treatment team consists of a physician, a physiotherapist and a social service worker. The main goal for the team is to make a survey of the patient's situation, in which the biomedical tradition to make a diagnosis is replaced by a disability diagnosis, with systematically identification of barriers for return to work. The conclusion of the team will be followed by a targeted rehabilitation plan. Factors assessed to be the major cause of the reduced function at work will have priority in the following rehabilitation process. One of the team members will be responsible for the further process to follow the plan to help the patient back to work, in cooperation with the patient, the workplace, the general practitioner, and NAV.
  Other Names: ISIVET; visual educational tool; interdisciplinary structured interview; multidisciplinary intervention; multidisciplinary treatment
  Arms: Intervention group
Behavioral: Control Group, Brief Intervention — The brief intervention is a standardized intervention and the essential features are interview and examination by a specialist in physical medicine and rehabilitation. Patients will be given time to express their concerns and problems in daily activities. The examination is thorough with detailed feedback on findings and normal functions, and clear and consistent explanations on pain and defense mechanisms. Somatic findings will be explained.Unless pathological findings, the patient will be encouraged to physical activity.
  Arms: Controll group

SUMMARY:
Musculoskeletal pain is very common in the normal population, and the reason for about 50 % of the long term sickness absence in Norway. Most of these patients have common, but troublesome subjective health complaints where pathological findings are absent or substantially less than expected compared to the reported intensity of the complaints. Psychosocial factors are important in the development of chronic complaints. In a large meta-analysis job satisfaction was found to be associated with mental health and subjective physical health. Individual factors are also important. Uncertainty related to the understanding of pain mechanisms, treatment strategies and management contribute to the problem.

Among patients sicklisted for musculoskeletal complaints, low back pain is the largest diagnose group. Most of these patients also have many other complaints. Previous studies have shown that for low back pain patients a brief intervention at a spine clinic with examination, information, reassurance, and encouragement to engage in physical activity as normal as possible, had significant effect in reducing sick leave. Other studies have shown that multidisciplinary rehabilitation for chronic low back pain has effect on sick leave. A Danish study from Arbeidsmiljøinstituttet report that interdisciplinary treatment for patients sicklisted for musculoskeletal complaints, had effect on socio-economic costs, pain, and function.

A treatment team consisting of various professionals is expensive, and in this study we will compare the simple, standardized brief intervention model with the more resource demanding interdisciplinary treatment for patients sicklisted for musculoskeletal complaints.

Research question / hypothesis: An interdisciplinary treatment model for musculoskeletal complaints - is it beneficial for reducing sickness absence?

DETAILED DESCRIPTION:
In 2007 The Government in Norway raised a fund to support efforts to reduce sickness absence, called "Raskere tilbake prosjekt". Helse Sør-Øst was invited to establish projects within their health care system, and the department of physical medicine and rehabilitation at Sykehuset Innlandet HF was assigned the task to constitute an outpatient-clinic for musculoskeletal diseases.

This initiative opened possibilities to explore new strategies based on science and own clinical experience to help these patients back to work without being confined to the traditional diagnose related examination and treatment offered in most clinics. In this project the main focus is directed towards work and barriers for working life. Because sickness absence often is multicausal and needs a bio-psycho-social approach, this should be reflected in the composition of the treatment team.

There is a great demand to make out how complex bio-psycho-social problems can be solved, organized, implemented, and have economic gains for the society. To answer these questions we need randomized controlled clinical studies, and we need documentation when new treatment models are offered to this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Musculoskeletal diagnosis
* Minimum 50% sick leave from work for not more than one year
* Minimum 50 % employed

Exclusion Criteria:

* Not sicklisted
* Sicklisted less than 50%
* Sicklisted > 1 year
* Less than 50% employed
* Pregnancy
* Does not speak Norwegian
* Psychiatric disease
* Osteoporosis
* Cancer disease
* Rheumatic disease
* Ongoing Insurance Compensation Case

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 284 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Sickness leave 1 year after inclusion | At 12 months after baseline
  In addition to the main outcome we will also evaluate job satisfaction, social support, coping, defense mechanisms, illness perception, function level, activity of daily living, psychological distress, and health complaints/pain as recorded by the questionnaires at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Eli M. Hagen, MD, PhD, Study Chair — Sykehuset Innlandet HF
Locations (1):
- Dep. of Physica. Medicin and Rehabilitation, Innlandet Hospital Trust, Ottestad, Ottestad, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brendbekken R, Eriksen HR, Grasdal A, Harris A, Hagen EM, Tangen T. Return to Work in Patients with Chronic Musculoskeletal Pain: Multidisciplinary Intervention Versus Brief Intervention: A Randomized Clinical Trial. J Occup Rehabil. 2017 Mar;27(1):82-91. doi: 10.1007/s10926-016-9634-5. PMID 26910406
- See also: Info about the project: Raskere tilbake — http://sykehuset-innlandet.no